CLINICAL TRIAL: NCT04738695
Title: SARS-CoV-2 Seroprevalence Among Nursing Home Staff and Residents in Belgium
Brief Title: SARS-CoV-2 Seroprevalence Among Nursing Home Staff and Residents (COVID-19)
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Collaborators: KU Leuven (Other); University of Liege (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08719
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: Covid19; SARS-CoV-2 Infection; Seroprevalence; Nursing home
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Capillary blood (whole blood) samples:
  * collection using point-of-care rapid SARS-CoV-2 antibody test
  * collection on Dry Blood Spot saver card
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing home residents/staff members: Follow-up of seroprevalence
  Interventions: Diagnostic Test: Point-of-care rapid anti-SARS-CoV-2 antibody test (Orient Gene Biotech) and Dry Blood Spot collection (Euroimmun)

INTERVENTIONS:
Diagnostic Test: Point-of-care rapid anti-SARS-CoV-2 antibody test (Orient Gene Biotech) and Dry Blood Spot collection (Euroimmun) — Bimonthly finger pricks with collection of 1-10 drops of capillary blood for detection of anti-SARS-CoV-2 immune markers

SUMMARY:
Assessment of the seroprevalence and sero-incidence of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) among Nursing Home (NH) residents and staff in Belgium.

DETAILED DESCRIPTION:
In this longitudinal cohort study, 3036, nursing home (NH) residents (1656) and staff (1380), spread over 69 nursing homes throughout Belgium will be repeatedly sampled at a 2-month interval. Seroprevalence and -incidence will be assessed by means of a point-of-care rapid antibody test with additional collection of a Dry Blood Spot sample for quantitative detection of immune markers*. Sample collection (capillary blood samples) at baseline (day 0, week 0) will start in a staggered way, so all baseline samples among the different nursing homes are collected within the first 21 days after collection of the first sample. Follow-up sample collection will occur with a 2-month interval in week 8, week 16, week 24, week 32 and week 40 after the baseline collection of that specific nursing home. At each timepoint, questionnaires will be taken concerning medical history, clinical outcomes and potential COVID-19 riskfactors. The recruited NHs will be equally spread across the Belgian territory according to geographic and demographic characteristics to guarantee general representativity. Forty-four participants (20 staff, 24 residents) will be randomly included per nursing home. (* collection of the Dry Blood Spot is part of a sub-study by Ghent University)

ELIGIBILITY:
Inclusion Criteria:

* residents and staff from Belgian nursing homes

Exclusion Criteria:

* service flat residents
* temporary staff, employed for a period of less then 1 year starting from baseline collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing Home residents and staff members.
Sampling Method: Probability Sample
Enrollment: 3008 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of seroprevalence of anti-SARS-CoV-2 antibodies among nursing home residents and staff in Belgium | "Month 0", "Month 2", "Month 4", "Month 6", "Month 8", "Month 10", "Month 13", "Month 16", "Month 19", "Month 22"
  Change of seroprevalence of anti-SARS-CoV-2 antibodies among Belgian nursing home residents and staff detected in their capillary blood by a point of care test during a period of 10 months.
Change in SARS-CoV-2 seroconversion among nursing home residents and staff in Belgium | "Month 0", "Month 2", "Month 4", "Month 6", "Month 8", "Month 10", "Month 13", "Month 16", "Month 19", "Month 22"
  Change in SARS-CoV-2 seroconversion among Belgian nursing home residents and staff conducted by detecting specific SARS-CoV-2 IgG/IgM in their capillary blood by a point of care test at each of the study follow-up testing points.

SECONDARY OUTCOMES:
Assess the risk of getting symptomatically SARS-CoV-2 infected between the seropositive and seronegative group at baseline | 10 months
  For all participants, the hazard of new symptomatic SARS-CoV-2 infections between sero-positive and -negative participants at the baseline visit will be estimated and reported as cumulative survival rates after 10 months of follow-up with 95% Confidence Interval (CI). The analysis will account the clustered nature of participants within NH and will be adjusted for the stratification factors province and type of participant (staff vs resident). If a vaccine would become available during the study period, the admission of a vaccine will be added as a time-varying covariate to the analysis.
Assess the proportion of deaths within 10 months between sero-positive and -negative participants at baseline visit for NH residents. | 10 months
  For NH residents, the proportion of deaths within 10 months of follow-up between sero-positive and -negative participants at the baseline visit will be assessed. Province, age, gender, care profile, presence of COVID-specific comorbidities at baseline and timevarying covariate COVID-19 vaccine will be considered for model adjustment.
Assess the seroconversion time in the group of sero-negative participants at baseline visit in relation to observed risk factors such as care dependency scale (for NH residents),type of job assignment and flu vaccination (for staff) | 10 months
  The sero-conversion time in the group of sero-negative participants at the baseline visit will be modelled separately for residents and staff, on the one hand assessing potential differences between care profiles or residence ward (dementia unit or not) for NH residents, and differences between flu vaccination status and type of job assignment for the staff on the other hand. For both types of participants the model will be adjusted for province, age, gender, presence of COVID-specific comorbidities at baseline and time-varying covariate COVID-19 vaccine.
Assess the duration of SARS-CoV-2 antigen specific seropositivity among NH residents and staff in Belgium. | 10 months
  The duration of SARS-CoV-2 antigen specific seropositivity among NH residents and staff in Belgium will be modelled by means of interval-censored survival analysis.
Assess the time until death within 10 months between sero-positive and -negative participants at baseline visit for NH residents | 10 months
  For NH residents, the time until death between sero-positive and -negative participants at the baseline visit will be assessed within 10 months. Province, age, gender, care profile, presence of COVID-specific comorbidities at baseline and timevarying covariate COVID-19 vaccine will be considered for model adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: An De Sutter, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request.
Supporting Information: Study Protocol, ICF
Time Frame: At the earliest 3 months after database lock, available for 10 years.
Access Criteria: Available on request through e-mail correspondence to principal investigator.

REFERENCES:
- [Background] Lipsitch M, Swerdlow DL, Finelli L. Defining the Epidemiology of Covid-19 - Studies Needed. N Engl J Med. 2020 Mar 26;382(13):1194-1196. doi: 10.1056/NEJMp2002125. Epub 2020 Feb 19. No abstract available. PMID 32074416
- [Derived] Meyers E, De Rop L, Deschepper E, Duysburgh E, De Burghgraeve T, Van Ngoc P, Digregorio M, Coen A, De Clercq N, Wallaert S, Buret L, Coenen S, De Sutter A, Scholtes B, Verbakel JY, Cools P, Heytens S. SARS-CoV-2 seroreversion and all-cause mortality in nursing home residents and staff post-primary course vaccination in Belgium between February and December 2021. Vaccine. 2025 Apr 2;51:126865. doi: 10.1016/j.vaccine.2025.126865. Epub 2025 Feb 20. PMID 39983537
- [Derived] Meyers E, De Rop L, Deschepper E, Duysburgh E, De Burghgraeve T, Van Ngoc P, Digregorio M, Delogne S, Coen A, De Clercq N, Buret L, Coenen S, De Sutter A, Scholtes B, Verbakel JY, Cools P, Heytens S. Prevalence of SARS-CoV-2 antibodies among Belgian nursing home residents and staff during the primary COVID-19 vaccination campaign. Eur J Gen Pract. 2023 Dec;29(2):2149732. doi: 10.1080/13814788.2022.2149732. Epub 2022 Nov 28. PMID 36440533